CLINICAL TRIAL: NCT02200107
Title: Implementing and Evaluating Integrated Medical and Physiotherapy Treatment Program for Osteoarthritis of the Knee by Family Doctors in Primary Care Clinics
Brief Title: Integrated Treatment Program for Osteoarthritis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OA-knee 015/2014
Record Dates: First submitted 2014-07-17; First posted 2014-07-25 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis Knee
Keywords: Osteoarthritis Knee; Self Care; Treatment Outcome; Patient Education as Topic; Physical Therapy Modalities
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (2):
- self management education (Experimental): self management education program delivered by family doctor in primary care clinics and during and physical therapy design
  Interventions: Behavioral: self management education
- control (No Intervention): Routine follow up according to standard practice

INTERVENTIONS:
Behavioral: self management education
  Arms: self management education

SUMMARY:
The purpose of this study is to determine the ability to assimilate and implement an integrated treatment program osteoarthritis of the knee, including the diagnosis and follow-up by a family physician in primary care clinics, combined with patient self-care training and physiotherapy program

ELIGIBILITY:
Inclusion Criteria:

* Active complaint of knee pain
* Diagnosis of knee osteoarthritis according to X-ray
* Morning stiffness of less than 30 minutes AND/OR crepitus in active movement
* Ability to read Hebrew

Exclusion Criteria:

* Previous participation in physiotherapy treatment program
* Gout in knee, rheumatoid arthritis, fibromyalgia
* Complaints that appear in a knee which was operated in the past
* Dementia
* Severe limitations in mobility

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in WOMAC ( Western Ontario and McMaster Universities Arthritis Index ) score during participating in the program | 0, 6 weeks, for intervention group after completing physical therapy program, for the control group after 6 months
  WOMAC score will be evaluated through a questionnaire (validated to Hebrew) at baseline and after a constant time period. For both groups (intervention and control) after 6 weeks from enrollment and then for the control group after 6 months, and for the intervention group after completing physical therapy program. we will assess the change from baseline.

SECONDARY OUTCOMES:
Change in VAS pain score during participating in the program | 0, 6 weeks, for intervention group after completing physical therapy program, for the control group after 6 months
  VAS score will be evaluated through a questionnaire (validated to Hebrew) at baseline and after a constant time period. For both groups (intervention and control) after 6 weeks from enrollment and then for the control group after 6 months, and for the intervention group after completing physical therapy program. we will assess the change from baseline.
Change in the consumption of drugs during participating in the program | 0, 6 weeks, for intervention group after completing physical therapy program, for the control group after 6 months
  Prescriptions given by family doctor, for treating patient's knee complaints. It will be evaluated by the medical record registration of the patients, at baseline and after a constant time period. For both groups (intervention and control) after 6 weeks from enrollment and then for the control group after 6 months, and for the intervention group after completing physical therapy program.
Changes in Referrals to specialists doctors during participating in the program | after 6 weeks since enrollment, and then for intervention group after completing physical therapy program, and for the control group after 6 months
  Referrals given by family doctor. It will be evaluated by the medical record registration of the patients, for both groups (intervention and control) after 6 weeks from enrollment and then for the control group after 6 months, and for the intervention group after completing physical therapy program.

OTHER OUTCOMES:
Patient satisfaction with treatment | 6 months after enrollment
  Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Avny, MD, Study Chair — Clalit Health Service
Locations (1):
- Clalit Health Service, Jerusalem, Israel